CLINICAL TRIAL: NCT03673943
Title: An Open-label, Single-dose, Single Arm, Single-center Clinical Trial of 64Cu(Copper)-DOTATATE (NETMedix™) PET-CT Scan for Imaging Patients With Known or Suspected Somatostatin Receptor-positive Neuroendocrine Tumors (NETs)
Brief Title: Imaging of Patients With Known or Suspected Somatostatin Receptor Positive Neuroendocrine Tumors Using Cu64-DOTATATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiomedix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 131797
Record Dates: First submitted 2018-08-23; First posted 2018-09-17 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 64Cu-DOTATATE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT imaging with 64Cu-DOTATATE (Experimental): 64Cu-DOTATATE is an investigational radioactive drug that binds to somatostatin receptors on neuroendocrine cancer cells.
  Interventions: Drug: 64Cu-DOTATATE

INTERVENTIONS:
Drug: 64Cu-DOTATATE — Detection of somatostatin positive lesions in NET
  Other Names: NETMEDIX

SUMMARY:
This is an open-label, single-dose, single-arm, single-center imaging study using DOTATATE peptide, labelled with the 64Cu tracer.

DETAILED DESCRIPTION:
In total, 59 subjects will be recruited in the study. The study will recruit both healthy volunteers as well as patients with confirmed or suspicious NET disease by histology or conventional anatomical and functional imaging modalities including but not limited to magnetic resonance imaging (MRI), and/or computed tomography (CT), and/or, F-18 FDG fluorodeoxyglucose PET (positron emission tomography)/CT and /or F-18 NaF sodium fluoride bone PET/CT and/or bone scintigraphy, and/or Octreoscan.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspicion of NET based on histology/ biopsy report.
* Confirmed or suspicion of NET based on conventional imaging scans of affected area such as MRI and/or contrast enhanced CT and/or an FDG PET
* CT scan and/or NaF PET-CT scan and/or OctreoScan® performed within 8 weeks prior to study date.

Exclusion Criteria:

* Pregnant, planning to be pregnant within the next two weeks
* Inability to provide written consent.
* Therapeutic use of any somatostatin analogue, including Sandostatin® long-acting and Lanreotide (within 28 days) and Sandostatin® (within 2 days) prior to study imaging. If a subject is on Sandostatin® long-acting or Lanreotide, a wash-out period of 28 days is required before the injection of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S Delpassand, MD, Study Director — Radiomedix, Inc.
Locations (1):
- Excel Diagnostics and Nuclear Oncology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delpassand ES, Ranganathan D, Wagh N, Shafie A, Gaber A, Abbasi A, Kjaer A, Tworowska I, Nunez R. 64Cu-DOTATATE PET/CT for Imaging Patients with Known or Suspected Somatostatin Receptor-Positive Neuroendocrine Tumors: Results of the First U.S. Prospective, Reader-Masked Clinical Trial. J Nucl Med. 2020 Jun;61(6):890-896. doi: 10.2967/jnumed.119.236091. Epub 2020 Jan 10. PMID 31924723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of Subjects (planned and analyzed): 63 Analyzed: In total, 63 subjects (59 from the Phase 3 study and 4 from the Phase 1 study) were injected with study drug at an intended dose of 4.0 mCi and met the criteria to be analyzed for safety and efficacy.
Groups:
- PET/CT Imaging With 64Cu-DOTATATE: 64Cu-DOTATATE is an investigational radioactive drug that binds to somatostatin receptors on NETs cancer cells.
  64Cu-DOTATATE: Detection of somatostin positive lesions in NET
Period: Overall Study
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The following analysis populations were defined: Efficacy Evaluable (EE) Population - consisted of all subjects who were enrolled in the study had an established SOT, were injected with 64Cu DOTATATE, and had an image read result using 64Cu-DOTATATE by three independent readers.
  Safety Population - The safety population consisted of all subjects who were enrolled in the study
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 54.37 (15.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of 64Cu-DOTATATE PET-CT Imaging for Detection of Somatostatin Receptor Positive SSTR (+) Tumor
Description: The number of patients with NETs disease that was confirmed by SSTR(+) imaging using 64Cu-DOTATATE PET/CT and In111-Octreoscan (considered as the standard of truth imaging) A total of 63 subjects have been enrolled in the studies; among them 42 patients with known or suspected NET based on histology, or conventional imaging, or clinical evaluations and 21 healthy volunteers.
Time Frame: 12 months
Population: The number of patients with SSTR(+) NETs identified using 64Cu-DOTATATE PET-CT imaging as well as by the standard of truth methods.
  A total of 63 subjects have been enrolled in the studies, including 42 patients with known or suspected NET based on histology, conventional imaging, or clinical evaluations and 21 healthy volunteers.
Measure: Count of Participants; unit: Participants
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
Number analyzed (Participants) | 62
Participants
  true positive | 30
  false negative | 3

2. Primary Outcome: Specificity of 64Cu- DOTATATE PET/CT Imaging for Detection of Neuroendocrine Tumor
Description: The number of subjects who have no SSTR (+) NETs as determined by 64Cu-DOTATATE PET/CT as well using the standard of truth imaging (In111-Octrescan SPECT/CT).
Time Frame: 12 months
Population: The specificity of 64Cu-DOTATATE imaging has defined the ability of a radiotracer to correctly identify subjects who do not have a disease. It is defined by number of subjects who had no SSTR(+) NETs based on 64Cu-DOTATATE PET/CT imaging as well as SOT imaging using In111-Octreoscan.
Measure: Count of Participants; unit: Participants
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
Number analyzed (Participants) | 62
Participants
  true negative | 28
  false positive | 1

3. Secondary Outcome: Detection of Localized or Metastatic SSTR Positive NETs Lesions Using Both 64Cu-DOTATATE PET/CT and Standard of Truth Imaging
Description: The number of patients with localized NETs or metastatic SSTR(+) neuroendocrine tumors that were detected by both 64Cu-DOTATATE and SOT
Time Frame: 12 months
Population: A number of subjects with localized SSTR(+) NETs or metastatic NETs detected by both Cu64-DOTATATE and SOT
Measure: Count of Participants; unit: Participants
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
Number analyzed (Participants) | 30
Participants
  localized NETs true positive | 2
  localized NEts false negative | 0
  metastatic NETs false positive | 0
  metastatic NETs true negative | 28

ADVERSE EVENTS:
Time Frame: Any adverse events observed or reported were recorded for up to 48 hours following study drug administration. In addition, observed or patient reported immediate adverse events including but not limited to pain, injection site reaction, headache, nausea, vomiting, flushing or other as reported, were assessed within 1 hour before and within 2 hours after the study drug administration
Arm/Group | PET/CT Imaging With 64Cu-DOTATATE
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 5/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/CT Imaging With 64Cu-DOTATATE (N=63)
nausea (grade 1) (Gastrointestinal disorders) | 1 (1) — All adverse events were either mild or moderate in severity. There were no adverse events that were severe, life-threatening or disabling, or that resulted in death. Adverse events that were mild in severity included nausea, vomiting, headache
headache (grade 1) (General disorders) | 1 (1)
syncope (grade 2) (General disorders) | 1 (1)
melanoderma (grade 1) (General disorders) | 1 (1)
flushing (grade 1) (General disorders) | 1 (1)
vomiting (both grade 1) (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT03673943/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT03673943/SAP_001.pdf